CLINICAL TRIAL: NCT03433417
Title: A Single-center, Prospective, Non-randomized, Open-label Clinical Study to Evaluate the Performance of the truSculpt Radiofrequency Device for Non-invasive Fat Reduction in Abdominal Tissue in Subjects Who Are Scheduled for Abdominoplasty
Brief Title: Performance Evaluation of the truSculpt Radiofrequency Device for Lipolysis of Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: C-17-TS13
Record Dates: First submitted 2018-02-05; First posted 2018-02-14 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Body Fat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Side (Experimental): One truSculpt treatment
  Interventions: Device: Cutera truSculpt
- Control Side (No Intervention): Untreated contralateral control

INTERVENTIONS:
Device: Cutera truSculpt — One truSculpt treatment delivered 0 to 90 days before scheduled Abdominoplasty to one side of the tissue to be removed during abdominoplasty
  Arms: Treatment Side

SUMMARY:
Clinical Study to Evaluate the Performance the truSculpt Radiofrequency Device for Lipolysis of Abdominal Fat

DETAILED DESCRIPTION:
A single-center, prospective, non-randomized, open-label study to evaluate the truSculpt Radiofrequency Device for non-invasive fat reduction in abdominal tissue for up to 14 subjects. Measurement will be histological evaluation of tissue for selective fat necrosis, with sparing of the dermis and epidermis, following truSculpt treatment vs. untreated contralateral control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 24 to 60 years of age (inclusive)
2. Fitzpatrick Skin Type I - VI (Appendix 3)
3. Has visible fat bulges or skin laxity in the abdominal region
4. Scheduled to undergo surgery (abdominoplasty).
5. Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.
6. Subject must agree to not undergo any other procedure(s) in the abdominal region during the study period.
7. Subject must be able to read, understand and sign the Informed Consent Form.
8. Subject must adhere to the follow-up schedule and study instructions.
9. Subject must adhere to the same diet/ exercise/medication regimen for the entire course of the study.
10. Willing to provide histology samples during the surgery from the intended to be harvested areas.
11. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug in the target area during the study period.
2. Any type of prior cosmetic treatment to the target area within 12 months of study participation e.g., radiofrequency, cryolysis or light-based treatments.
3. Any prior invasive cosmetic surgery to the target area, such as liposuction.
4. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.
5. Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.
6. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.
7. Diagnosed or documented immune system disorders.
8. History of any disease or condition that could impair wound healing.
9. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.
10. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing in the treatment area.
11. Infection, dermatitis, rash or other skin abnormality in the target area.
12. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.
13. Pregnant or currently breastfeeding.
14. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Cutera Research Center
Locations (1):
- Cutera Research Center, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: abdominal subareas
Groups:
- All Study Participants: One truSculpt treatment will be performed before scheduled Abdominoplasty on one abdominal subarea. The other bilateral abdominal subarea will not be treated and act as a control.
  Two biopsies will be harvested from tissue removed during the Abdominoplasy: one from the treated area and one from the control area.
Period: Overall Study
Arm/Group | All Study Participants
Started | 12; 24 abdominal subareas
Treatment With TruSculpt Device | 12; 12 abdominal subareas
No Treatment With TruSculpt Device | 12; 12 abdominal subareas
Completed | 12; 24 abdominal subareas
Not Completed | 0; 0 abdominal subareas

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: One truSculpt treatment
  Cutera truSculpt: one truSculpt treatment before scheduled Abdominoplasty on tissue to be removed during abdominoplasty
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who's Abdominal Tissue Showed Necrosis or Inflammatory Immune Cell Response
Description: Descriptive histological evaluation of abdominal tissue for selective fat necrosis, with sparing of the dermis and epidermis, following one truSculpt treatment vs. untreated bilateral control. A responder is a biopsy sample that shows necrosis or inflammatory immune cell response.
Time Frame: 0 to 90 days
Population: 24 biopsy samples were collected; however, the treatment side and untreated bilateral control side biopsy samples from 1 participant were lost during transit to the histology lab.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants - Treatment Side: Biopsy sample of abdominal tissue taken immediately prior to participant's scheduled abdominoplasty from the side that received one truSculpt RF treatment 0 to 90 days prior to the scheduled abdominoplasty.
- All Study Participants - Untreated Bilateral Control Side: Biopsy sample of abdominal tissue taken immediately prior to participant's scheduled abdominoplasty from the untreated bilateral control side.
Arm/Group | All Study Participants - Treatment Side | All Study Participants - Untreated Bilateral Control Side
Number analyzed (Participants) | 11 | 11
Participants | 10 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Treatment Side | Control Side
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Side (N=12) | Control Side (N=12)
Erythema (Skin and subcutaneous tissue disorders) | 12 (12) | 0
Edema (Skin and subcutaneous tissue disorders) | 12 (12) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03433417/Prot_SAP_000.pdf